CLINICAL TRIAL: NCT05828043
Title: Brain Aging: Muscle-to-brain Axis Modulates Physio-cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Liang-Kung Chen,MD, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YM109161F
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Age-related Cognitive Decline; Age-related Physiology Decline
Keywords: frailty; cognitive impairment; physio-cognitive decline syndrome; dementia; biomarkers; skeletal muscle; aging; neuroimaging; multidomain intervention
MeSH Terms: conditions — Frailty; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care group (No Intervention): Provide conventional health educations in every three-month interval
- Multidomain intervention group (Experimental): The multidomain intervention program is designed as structural training sessions of 2-hour training sessions two times per week.
  Interventions: Behavioral: Multi-domain intervention

INTERVENTIONS:
Behavioral: Multi-domain intervention — Each session comprises of 45 minutes physical fitness activities targeting on muscle strength, balance, and flexibility; 1-hour cognitive training primarily on reasoning and memory exercises; and 15-minute for nutritional advices based on national diet guidelines for older adults
  Arms: Multidomain intervention group

SUMMARY:
The primary goal is to develop a multidomain intervention program focused on preserving global or regional brain volume and functions while simultaneously improving physical mobility and cognitive functions in older individuals with mobility frailty. This initiative seeks to unravel the brain-muscle axis mechanisms contributing to the accelerated functional declines observed in older populations. Moreover, our objective includes examining the relationships between the intervention and a broad spectrum of clinical characteristics, phenotypic traits, biochemical profiles, myokines, proteomics, metabolomics, brain imaging, and our previously identified discoveries involving exosomal miRNA.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of 12-month multidomain intervention program among community-living older adults with early physical or cognitive impairments.

Inclusion criteria are: (1) community-dwelling adults aged ≥ 65 years, (2) slow gait speed (<1 m/s in 6-meter walk test) or weakness (dominant handgrip strength <28 kg in men, <18 kg in women); subjects with the following conditions will be excluded: (1) established diagnosis of dementia, Parkinsonism or other neurodegenerative disease (2) disable status: mobility-limiting conditions, (3) active, acute diseases receiving treatment, such as cancer, heart failure, COPD and so on, (4) estimated life expectancy <12 months, (5) current nursing home residents.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65 years
* slow gait speed (<1 m/s in 6-meter walk test) or weakness (dominant handgrip strength <28 kg in men, <18 kg in women)

Exclusion Criteria:

* established diagnosis of dementia, Parkinsonism or other mobility-limiting, disable conditions
* active, acute diseases receiving treatment, such as cancer, heart failure, COPD and so on
* estimated life expectancy <12 months
* current nursing home residents

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change in brain structures on MRI | baseline, 12 month
  Change in brain structures from baseline to 12 months in all participants
Change in Physical performance | baseline, 6, 12 month
  Change in hand-grip strength (kg), six-meter walking speed (m/s), and 5 times sit to stand test from baseline to 12 months in all participants

SECONDARY OUTCOMES:
Life quality SF12 | baseline, 6, 12 month
  measured by the 12-Item Short Form Health Survey (SF-12).
Change in Complete blood count | baseline, 6, 12 month
  Change in Complete blood count from baseline to 12 months in all participants
Change in Nutrition intake | baseline, 6, 12 month
  measured by Mini-nutritional assessment questionnaire. ranged 0-30, higher values represent a better condition
Change in depression | baseline, 6, 12 month
  measured by the Center for Epidemiological Studies-Depression (CES-D) ranged 0-60, higher values represent a worse condition
Change in cognitive ability | baseline, 6, 12 month
  Change in cognitive function measure by MoCA ranged 0-30, higher values represent a better condition
Change in International Physical Activity Questionnaire (IPAQ) | baseline, 6, 12 month
  Change in physical activity measured by IPAQ, indicates that spent being physically active than the prior 7 days.There are no established thresholds for presenting MET-minutes, the IPAQ Research Committee proposes that reported as comparisons of median values and interquartile ranges for different populations from baseline to 12 months in all participants. The higher values represent a better activity.
Change in Vitamin D3 25-OH | baseline, 6, 12 month
  Change in Vitamin D3 25-OH concentration from baseline to 12 months in all participants
Change in DHEA-S | baseline, 6, 12 month
  Change in DHEA-S concentration from baseline to 12 months in all participants
Change in IGF-1 | baseline, 6, 12 month
  Change in IGF-1 concentration from baseline to 12 months in all participants
Change in Homocysteine | baseline, 6, 12 month
  Change in Homocysteine concentration from baseline to 12 months in all participants
Change in hs-CRP | baseline, 6, 12 month
  Change in hs-CRP concentration from baseline to 12 months in all participants
Change in Zinc | baseline, 6, 12 month
  Change in Zinc concentration from baseline to 12 months in all participants
Change in TSH | baseline, 6, 12 month
  Change in TSH concentration from baseline to 12 months in all participants
Change in Myostatin | baseline, 6, 12 month
  Change in Myostatin concentration from baseline to 12 months in all participants
Change in Activing A | baseline, 6, 12 month
  Change in Activing A concentration from baseline to 12 months in all participants
Change in Follistatin | baseline, 6, 12 month
  Change in Follistatin concentration from baseline to 12 months in all participants
Change in Relative appendicular skeletal muscle index (RASM) | baseline, 6, 12 month
  Change in RASM from baseline to 12 months in all participants
Change in body fat % | baseline, 6, 12 month
  Change in body fat % from baseline to 12 months in all participants

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, M.D., PhD, Study Director — Center for Healthy Longevity and Aging Sciences, National Yang Ming Chiao Tung University
Locations (1):
- Center for Healthy Longevity and Aging Sciences, National Yang Ming Chiao Tung University, Taipei, Taiwan